CLINICAL TRIAL: NCT05732064
Title: Effects of Low-dose Dexmedetomidine-esketamine Combined Nasal Administration at Night on Perioperative Sleep Quality in Breast Cancer Patients: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Dexmedetomidine-esketamine Combined Nasal Administration and Perioperative Sleep Quality
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and chairman, Department of Anesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022-761
Record Dates: First submitted 2023-01-29; First posted 2023-02-16 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Perioperative Period; Dexmedetomidine; Esketamine; Sleep Quality
Keywords: Breast Cancer; Perioperative period; Dexmedetomidine; Esketamine; Sleep quality
MeSH Terms: conditions — Breast Neoplasms; Sleep Initiation and Maintenance Disorders | interventions — Dexmedetomidine; Esketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine and esketamine (Experimental): Dexmedetomidine 0.5 microgram/kg (300 microgram/ml) and esketamine 0.2 mg/kg (25 mg/ml) are administered via nasal cavity at 20:00 pm the day before surgery, the day of surgery, and the first day after surgery.
  Interventions: Drug: Dexmedetomidine; Drug: Esketamine
- Normal saline (Placebo Comparator): Same volumes of normal saline are administered via nasal cavity at 20:00 pm the day before surgery, the day of surgery, and the first day after surgery.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 0.5 microgram/kg (300 microgram/ml) is administered via nasal cavity at 20:00 pm the day before surgery, the day of surgery, and the first day after surgery.
  Arms: Dexmedetomidine and esketamine
Drug: Esketamine — Esketamine 0.2 mg/kg (25 mg/ml) is administered via nasal cavity at 20:00 pm the day before surgery, the day of surgery, and the first day after surgery.
  Arms: Dexmedetomidine and esketamine
Drug: Normal saline — Normal saline of same volume is administered via nasal cavity at 20:00 pm the day before surgery, the day of surgery, and the first day after surgery.
  Arms: Normal saline

SUMMARY:
Breast cancer patients often have sleep disturbances during the perioperative period. Dexmedetomidine is a highly selective alpha 2-adrenoceptor agonist with sedative, anxiolytic, and analgesic effects. Previous studies showed that night-time low-dose dexmedetomidine infusion improved sleep quality. Esketamine is a N-methyl-D-aspartic acid receptor antagonist and has been used as an anesthetic and analgesic. Recent studies showed that low-dose esketamine has anti-depressive and sleep-promoting effects. The investigators suppose that low-dose dexmedetomidine-esketamine combined nasal administration at night can improve perioperative sleep quality in patients scheduled for breast cancer surgery.

DETAILED DESCRIPTION:
Normal sleep is important for maintaining both physical and mental health. Patients who are scheduled for breast cancer surgery often have sleep disturbances during the perioperative period. Patients with persistent sleep disturbances have increased sensitivity to pain and are at increased risk of developing chronic postsurgical pain.

Dexmedetomidine is a highly selective alpha 2-adrenoceptor agonist with sedative, anxiolytic, and analgesic effects. Previous studies showed that night-time low-dose dexmedetomidine infusion improves sleep quality. Nasal administration of dexmedetomidine has been used in children as a premedication and in adults to reduce emergence agitation.

Esketamine is a N-methyl-D-aspartic acid receptor antagonist and has been used as an anesthetic and analgesic. Recent studies showed that low-dose esketamine has anti-depressive and sleep-promoting effects. Nasal administration of esketamine has been used in children to relieve pain and in adults for treatment-resistant depression.

This randomized trial is designed to test the hypothesis that combined nasal administration of low-dose dexmedetomidine-esketamine at night can improve perioperative sleep quality in patients scheduled for breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years or older;
* Diagnosed with breast cancer and scheduled for surgical resection;
* Signed the informed consent form.

Exclusion Criteria:

* Not suitable for nasal administration because of nasal cavity diseases (rhinitis, nasal polyps, or nasal membrane congestion by any reason);
* History of schizophrenia, epilepsy, Parkinson's disease, or myasthenia gravis;
* Unable to communicate due to coma, delirium, severe dementia, or language barrier before surgery;
* History of intracranial injury or neurosurgery;
* Taking sedative/hypnotics for sleep in the last month;
* Preoperative sleep apnea (diagnosed with sleep apnea, or at high risk of sleep apnea according to STOP-Bang assessment);
* History of hyperthyroidism and pheochromocytoma;
* Preoperative LVEF<30%; sick sinus syndrome, severe sinus bradycardia (heart rate<50 beats/min), or atrioventricular block of degree II or higher without pacemaker; use vasopressors with systolic blood pressure <90 mmHg;
* Severe liver dysfunction (Child-Pugh C classification), severe renal dysfunction (dialysis before surgery), or Amercian Society of Anesthesiologists classification ≥IV;
* Allergic to dexmedetomidine and/or esketamine, or other conditions that are considered unsuitable for study participation;
* Body mass index >30 kg/m2;
* Enrolled in other clinical studies.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-07-26 (Actual)

PRIMARY OUTCOMES:
Subjective sleep quality (the night of surgery) | The night on the day of surgery
  Subjective sleep quality is assessed with the Richards-Campbell Sleep Questionnaire (RCSQ). RCSQ is a self-reported measure that evaluated perception of nighttime sleep in five items, including sleep depth, sleep latency, number of awakenings, returning to sleep, and overall sleep quality. Each item was assessed with a 100-millimeter visual analog scale (score ranges from 0 to 100, with higher scores representing better sleep). The mean score of the five items represents the overall RCSQ score.

SECONDARY OUTCOMES:
Subjective sleep quality (the night before and the first night after surgery) | The night before surgery and the first night after surgery
  Subjective sleep quality if assessed with the RCSQ. RCQS is a self-reported measure that evaluated perception of nighttime sleep in five items, including sleep depth, sleep latency, number of awakenings, returning to sleep, and overall sleep quality. Each item was assessed with a 100-millimeter visual analog scale (score ranges from 0 to 100, with higher scores representing better sleep). The mean score of the five items represents the overall RCSQ score.
Objective sleep quality - total sleep time | The night before surgery, the night on the day of surgery, and the first night after surgery
  Objective sleep quality is assessed with the actigraphy.
Objective sleep quality - sleep efficiency | The night before surgery, the night on the day of surgery, and the first night after surgery
  Objective sleep quality is assessed with the actigraphy.
Objective sleep quality - sleep latency | The night before surgery, the night on the day of surgery, and the first night after surgery
  Objective sleep quality is assessed with the actigraphy.
Objective sleep quality - wake-up time after falling asleep | The night before surgery, the night on the day of surgery, and the first night after surgery
  Objective sleep quality is assessed with the actigraphy.
Intensity of acute pain | At 2 hours after surgery and twice daily during the first 2 postoperative days
  Intensity of acute pain is assessed with the numeric rating scale, an 11-point scale where 0=no pain and 10=the worst pain.
Subjective sleep quality at 30 days | At 30 days after surgery
  Subjective sleep quality at 30 days is assessed with the Pittsburgh Sleep Quality Index (PSQI). PSQI is a 7-item questionnaire consisting 19 self-rated questions that assesses sleep quality over the last month, each weighted equally on a 0-3 scale; higher scores indicate worse sleep quality.

OTHER OUTCOMES:
Use of supplemental analgesics | Within the first 2 days after surgery
  Include opioids and non-opioid analgesics.
Severity of anxiety | Before hospital discharge
  Anxiety is assessed with the Generalized Anxiexy Disorde-7 (GAD-7). GAD-7 contains 7 items assessing the core symptoms of anxiety. Patients rate their frequency of symptoms within the last two weeks on a four-point scale ranging from "not at all" to "almost every day". Scores range from 0 to 21, with higher scores indicating more severe anxiety.
Severity of depression | Before hospital discharge
  Depression is assessed with the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 includes 9-item requiring responses of 0 (not at all) to 3 (nearly every day) to assess the occurrence of depressive symptoms over the last two weeks. It has 8 items on depressive symptoms and 1 focused on suicidal ideation. Total scores range from 0 to 27, with higher score indicating more severe symptoms.
Length of hospital stay after surgery | Up to 30 days after surgery
  Length of hospital stay after surgery
Occurrence of postoperative complications | Up to 30 days after surgery
  Postoperative complications are defined as new-onset medical events that are deemed harmful and required therapeutic intervention, that is grade II or higher on the Clavien-Dindo classification.
Occurrence of Chronic Postoperative Pain | At 3 months after surgery
  Chronic Postoperative Pain (CPSP) is defined as pain persisted for at least three months after surgery, that was not present before surgery or that had different characteristics, and other possible causes of the pain were excluded (e.g., cancer recurrence, infection).
Severity of chronic pain | At 3 months after surgery
  Severity of chronic pain is assessed with the Brief Pain Inventory (BPI). The BPI gives two main scores: a pain severity score and a pain interference score. The pain severity score is calculated from the four items about pain intensity. Each item is rated from 0, no pain, to 10, pain as bad as you can imagine, and contributes with the same weight to the final score, ranging from 0 to 40.
Interference of chronic pain | At 3 months after surgery
  Interference of chronic pain is assessed with the Brief Pain Inventory (BPI). The BPI gives two main scores: a pain severity score and a pain interference score. The pain interference score corresponds to the item on pain interference. The seven subitems are rated from 0, does not interfere, to 10, completely interferes, and contributes with the same weight to the final score, ranging from 0 to 70.
Life quality assessed with the EORTC QLQ-BR53 (part of EORTC-C30) | At 3 months after surgery
  Quality of life is assessed with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Breast Cancer 53 (EORTC QLQ-BR53), including European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC-C30) and EORTC-BR23. EORTC QLQ-C30 contains 30 items (items 29 and 30 are classified into 7 degrees regarding to patients' response, scoring from 1 to 7; remaining items are divided into 4 degrees, including "Not at all", "A little", "Quite a bit", and "Very much", with a score from 1 to 4). All patient rated scores are linearly converted into a scale from 0 to 100 for analysis. Higher scores represent worse QoL on symptom aspects, whereas higher scores on functional interference correlate with better function.
Life quality assessed with the EORTC QLQ-BR53 (part of EORTC-BR23) | At 3 months after surgery
  Quality of life is assessed with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Breast Cancer 53 (EORTC QLQ-BR53), including European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC-C30) and EORTC-BR23. EORTC QLQ-BR23 contains 23 items. Each item used a 4-point Likert scale (i.e. "not at all", "a little", "quite a bit", and "very much"). All patient rated scores are linearly converted into a scale from 0 to 100 for analysis. Higher scores represent worse QoL on symptom aspects, whereas higher scores on functional interference correlate with better function.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijin, Bejing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sancho-Garnier H, Colonna M. [Breast cancer epidemiology]. Presse Med. 2019 Oct;48(10):1076-1084. doi: 10.1016/j.lpm.2019.09.022. Epub 2019 Nov 6. French. PMID 31706896
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Lei S, Zheng R, Zhang S, Wang S, Chen R, Sun K, Zeng H, Zhou J, Wei W. Global patterns of breast cancer incidence and mortality: A population-based cancer registry data analysis from 2000 to 2020. Cancer Commun (Lond). 2021 Nov;41(11):1183-1194. doi: 10.1002/cac2.12207. Epub 2021 Aug 16. PMID 34399040
- [Background] Bundred JR, Michael S, Stuart B, Cutress RI, Beckmann K, Holleczek B, Dahlstrom JE, Gath J, Dodwell D, Bundred NJ. Margin status and survival outcomes after breast cancer conservation surgery: prospectively registered systematic review and meta-analysis. BMJ. 2022 Sep 21;378:e070346. doi: 10.1136/bmj-2022-070346. PMID 36130770
- [Background] Tsaras K, Papathanasiou IV, Mitsi D, Veneti A, Kelesi M, Zyga S, Fradelos EC. Assessment of Depression and Anxiety in Breast Cancer Patients: Prevalence and Associated Factors. Asian Pac J Cancer Prev. 2018 Jun 25;19(6):1661-1669. doi: 10.22034/APJCP.2018.19.6.1661. PMID 29938451
- [Background] Carreira H, Williams R, Muller M, Harewood R, Stanway S, Bhaskaran K. Associations Between Breast Cancer Survivorship and Adverse Mental Health Outcomes: A Systematic Review. J Natl Cancer Inst. 2018 Dec 1;110(12):1311-1327. doi: 10.1093/jnci/djy177. PMID 30403799
- [Background] Kwak A, Jacobs J, Haggett D, Jimenez R, Peppercorn J. Evaluation and management of insomnia in women with breast cancer. Breast Cancer Res Treat. 2020 Jun;181(2):269-277. doi: 10.1007/s10549-020-05635-0. Epub 2020 Apr 20. PMID 32314110
- [Background] Fleming L, Randell K, Stewart E, Espie CA, Morrison DS, Lawless C, Paul J. Insomnia in breast cancer: a prospective observational study. Sleep. 2019 Mar 1;42(3):zsy245. doi: 10.1093/sleep/zsy245. PMID 30521041
- [Background] Siegel JM. Sleep viewed as a state of adaptive inactivity. Nat Rev Neurosci. 2009 Oct;10(10):747-53. doi: 10.1038/nrn2697. Epub 2009 Aug 5. PMID 19654581
- [Background] Hungs M. Fundamentals of sleep medicine [J]. JAMA, 2012, 307(12): 1320-1321.
- [Background] Mansano-Schlosser TC, Ceolim MF, Valerio TD. Poor sleep quality, depression and hope before breast cancer surgery. Appl Nurs Res. 2017 Apr;34:7-11. doi: 10.1016/j.apnr.2016.11.010. Epub 2016 Nov 17. PMID 28342628
- [Background] Su X, Wang DX. Improve postoperative sleep: what can we do? Curr Opin Anaesthesiol. 2018 Feb;31(1):83-88. doi: 10.1097/ACO.0000000000000538. PMID 29120927
- [Background] Fekih-Romdhane F, Achouri L, Hakiri A, Jaidane O, Rahal K, Cheour M. Hopelessness is associated with poor sleep quality after breast cancer surgery among Tunisian women. Curr Probl Cancer. 2020 Feb;44(1):100504. doi: 10.1016/j.currproblcancer.2019.100504. Epub 2019 Sep 17. PMID 31548046
- [Background] Shammas RL, Marks CE, Broadwater G, Le E, Glener AD, Sergesketter AR, Cason RW, Rezak KM, Phillips BT, Hollenbeck ST. The Effect of Lavender Oil on Perioperative Pain, Anxiety, Depression, and Sleep after Microvascular Breast Reconstruction: A Prospective, Single-Blinded, Randomized, Controlled Trial. J Reconstr Microsurg. 2021 Jul;37(6):530-540. doi: 10.1055/s-0041-1724465. Epub 2021 Feb 6. PMID 33548936
- [Background] Xie L, Kang H, Xu Q, Chen MJ, Liao Y, Thiyagarajan M, O'Donnell J, Christensen DJ, Nicholson C, Iliff JJ, Takano T, Deane R, Nedergaard M. Sleep drives metabolite clearance from the adult brain. Science. 2013 Oct 18;342(6156):373-7. doi: 10.1126/science.1241224. PMID 24136970
- [Background] Ratner V, Gao Y, Lee H, Elkin R, Nedergaard M, Benveniste H, Tannenbaum A. Cerebrospinal and interstitial fluid transport via the glymphatic pathway modeled by optimal mass transport. Neuroimage. 2017 May 15;152:530-537. doi: 10.1016/j.neuroimage.2017.03.021. Epub 2017 Mar 18. PMID 28323163
- [Background] Irwin MR. Sleep and inflammation: partners in sickness and in health. Nat Rev Immunol. 2019 Nov;19(11):702-715. doi: 10.1038/s41577-019-0190-z. PMID 31289370
- [Background] Yu J, Rawtaer I, Fam J, Jiang MJ, Feng L, Kua EH, Mahendran R. Sleep correlates of depression and anxiety in an elderly Asian population. Psychogeriatrics. 2016 May;16(3):191-5. doi: 10.1111/psyg.12138. Epub 2015 Jul 16. PMID 26179204
- [Background] Dzierzewski JM, Dautovich N, Ravyts S. Sleep and Cognition in Older Adults. Sleep Med Clin. 2018 Mar;13(1):93-106. doi: 10.1016/j.jsmc.2017.09.009. Epub 2017 Dec 8. PMID 29412987
- [Background] Fang H, Tu S, Sheng J, Shao A. Depression in sleep disturbance: A review on a bidirectional relationship, mechanisms and treatment. J Cell Mol Med. 2019 Apr;23(4):2324-2332. doi: 10.1111/jcmm.14170. Epub 2019 Feb 7. PMID 30734486
- [Background] Bubu OM, Brannick M, Mortimer J, Umasabor-Bubu O, Sebastiao YV, Wen Y, Schwartz S, Borenstein AR, Wu Y, Morgan D, Anderson WM. Sleep, Cognitive impairment, and Alzheimer's disease: A Systematic Review and Meta-Analysis. Sleep. 2017 Jan 1;40(1). doi: 10.1093/sleep/zsw032. PMID 28364458
- [Background] Mogavero MP, DelRosso LM, Fanfulla F, Bruni O, Ferri R. Sleep disorders and cancer: State of the art and future perspectives. Sleep Med Rev. 2021 Apr;56:101409. doi: 10.1016/j.smrv.2020.101409. Epub 2020 Nov 28. PMID 33333427
- [Background] Korostovtseva L, Bochkarev M, Sviryaev Y. Sleep and Cardiovascular Risk. Sleep Med Clin. 2021 Sep;16(3):485-497. doi: 10.1016/j.jsmc.2021.05.001. Epub 2021 Jun 25. PMID 34325825
- [Background] Hajj A, Hachem R, Khoury R, Hallit S, ElJEBBAWI B, Nasr F, El Karak F, Chahine G, Kattan J, Rabbaa Khabbaz L. Clinical and genetic factors associated with anxiety and depression in breast cancer patients: a cross-sectional study. BMC Cancer. 2021 Jul 30;21(1):872. doi: 10.1186/s12885-021-08615-9. PMID 34330229
- [Background] Civilotti C, Botto R, Maran DA, Leonardis B, Bianciotto B, Stanizzo MR. Anxiety and Depression in Women Newly Diagnosed with Breast Cancer and Waiting for Surgery: Prevalence and Associations with Socio-Demographic Variables. Medicina (Kaunas). 2021 May 7;57(5):454. doi: 10.3390/medicina57050454. PMID 34066935
- [Background] Nelson LE, Lu J, Guo T, Saper CB, Franks NP, Maze M. The alpha2-adrenoceptor agonist dexmedetomidine converges on an endogenous sleep-promoting pathway to exert its sedative effects. Anesthesiology. 2003 Feb;98(2):428-36. doi: 10.1097/00000542-200302000-00024. PMID 12552203
- [Background] Alexopoulou C, Kondili E, Diamantaki E, Psarologakis C, Kokkini S, Bolaki M, Georgopoulos D. Effects of dexmedetomidine on sleep quality in critically ill patients: a pilot study. Anesthesiology. 2014 Oct;121(4):801-7. doi: 10.1097/ALN.0000000000000361. PMID 24988068
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Zhang DF, Su X, Meng ZT, Li HL, Wang DX, Xue-Ying Li, Maze M, Ma D. Impact of Dexmedetomidine on Long-term Outcomes After Noncardiac Surgery in Elderly: 3-Year Follow-up of a Randomized Controlled Trial. Ann Surg. 2019 Aug;270(2):356-363. doi: 10.1097/SLA.0000000000002801. PMID 29742525
- [Background] Jun JH, Kim KN, Kim JY, Song SM. The effects of intranasal dexmedetomidine premedication in children: a systematic review and meta-analysis. Can J Anaesth. 2017 Sep;64(9):947-961. doi: 10.1007/s12630-017-0917-x. Epub 2017 Jun 21. PMID 28639236
- [Background] Li A, Yuen VM, Goulay-Dufay S, Sheng Y, Standing JF, Kwok PCL, Leung MKM, Leung AS, Wong ICK, Irwin MG. Pharmacokinetic and pharmacodynamic study of intranasal and intravenous dexmedetomidine. Br J Anaesth. 2018 May;120(5):960-968. doi: 10.1016/j.bja.2017.11.100. Epub 2018 Feb 2. PMID 29661413
- [Background] Uusalo P, Seppanen SM, Jarvisalo MJ. Feasibility of Intranasal Dexmedetomidine in Treatment of Postoperative Restlessness, Agitation, and Pain in Geriatric Orthopedic Patients. Drugs Aging. 2021 May;38(5):441-450. doi: 10.1007/s40266-021-00846-6. Epub 2021 Mar 16. PMID 33728561
- [Background] Barrett W, Buxhoeveden M, Dhillon S. Ketamine: a versatile tool for anesthesia and analgesia. Curr Opin Anaesthesiol. 2020 Oct;33(5):633-638. doi: 10.1097/ACO.0000000000000916. PMID 32826629
- [Background] Wolff K, Winstock AR. Ketamine : from medicine to misuse. CNS Drugs. 2006;20(3):199-218. doi: 10.2165/00023210-200620030-00003. PMID 16529526
- [Background] Feinberg I, Campbell IG. Ketamine administration during waking increases delta EEG intensity in rat sleep. Neuropsychopharmacology. 1993 Aug;9(1):41-8. doi: 10.1038/npp.1993.41. PMID 8397722
- [Background] Duncan WC, Sarasso S, Ferrarelli F, Selter J, Riedner BA, Hejazi NS, Yuan P, Brutsche N, Manji HK, Tononi G, Zarate CA. Concomitant BDNF and sleep slow wave changes indicate ketamine-induced plasticity in major depressive disorder. Int J Neuropsychopharmacol. 2013 Mar;16(2):301-11. doi: 10.1017/S1461145712000545. Epub 2012 Jun 7. PMID 22676966
- [Background] Faraguna U, Vyazovskiy VV, Nelson AB, Tononi G, Cirelli C. A causal role for brain-derived neurotrophic factor in the homeostatic regulation of sleep. J Neurosci. 2008 Apr 9;28(15):4088-95. doi: 10.1523/JNEUROSCI.5510-07.2008. PMID 18400908
- [Background] Song B, Zhu J. A Novel Application of Ketamine for Improving Perioperative Sleep Disturbances. Nat Sci Sleep. 2021 Dec 25;13:2251-2266. doi: 10.2147/NSS.S341161. eCollection 2021. PMID 34992482
- [Background] Duncan WC Jr, Ballard ED, Zarate CA. Ketamine-Induced Glutamatergic Mechanisms of Sleep and Wakefulness: Insights for Developing Novel Treatments for Disturbed Sleep and Mood. Handb Exp Pharmacol. 2019;253:337-358. doi: 10.1007/164_2017_51. PMID 28939975
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Abdallah CG, Adams TG, Kelmendi B, Esterlis I, Sanacora G, Krystal JH. KETAMINE'S MECHANISM OF ACTION: A PATH TO RAPID-ACTING ANTIDEPRESSANTS. Depress Anxiety. 2016 Aug;33(8):689-97. doi: 10.1002/da.22501. Epub 2016 Apr 6. PMID 27062302
- [Background] Newport DJ, Carpenter LL, McDonald WM, Potash JB, Tohen M, Nemeroff CB; APA Council of Research Task Force on Novel Biomarkers and Treatments. Ketamine and Other NMDA Antagonists: Early Clinical Trials and Possible Mechanisms in Depression. Am J Psychiatry. 2015 Oct;172(10):950-66. doi: 10.1176/appi.ajp.2015.15040465. PMID 26423481
- [Background] Kishimoto T, Chawla JM, Hagi K, Zarate CA, Kane JM, Bauer M, Correll CU. Single-dose infusion ketamine and non-ketamine N-methyl-d-aspartate receptor antagonists for unipolar and bipolar depression: a meta-analysis of efficacy, safety and time trajectories. Psychol Med. 2016 May;46(7):1459-72. doi: 10.1017/S0033291716000064. Epub 2016 Feb 12. PMID 26867988
- [Background] Bartova L, Papageorgiou K, Milenkovic I, Dold M, Weidenauer A, Willeit M, Winkler D, Kasper S. Rapid antidepressant effect of S-ketamine in schizophrenia. Eur Neuropsychopharmacol. 2018 Aug;28(8):980-982. doi: 10.1016/j.euroneuro.2018.05.007. Epub 2018 Jul 2. PMID 30041987
- [Background] Molero P, Ramos-Quiroga JA, Martin-Santos R, Calvo-Sanchez E, Gutierrez-Rojas L, Meana JJ. Antidepressant Efficacy and Tolerability of Ketamine and Esketamine: A Critical Review. CNS Drugs. 2018 May;32(5):411-420. doi: 10.1007/s40263-018-0519-3. PMID 29736744
- [Background] Canuso CM, Singh JB, Fedgchin M, Alphs L, Lane R, Lim P, Pinter C, Hough D, Sanacora G, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine for the Rapid Reduction of Symptoms of Depression and Suicidality in Patients at Imminent Risk for Suicide: Results of a Double-Blind, Randomized, Placebo-Controlled Study. Am J Psychiatry. 2018 Jul 1;175(7):620-630. doi: 10.1176/appi.ajp.2018.17060720. Epub 2018 Apr 16. PMID 29656663
- [Background] Segmiller F, Ruther T, Linhardt A, Padberg F, Berger M, Pogarell O, Moller HJ, Kohler C, Schule C. Repeated S-ketamine infusions in therapy resistant depression: a case series. J Clin Pharmacol. 2013 Sep;53(9):996-8. doi: 10.1002/jcph.122. Epub 2013 Jul 24. No abstract available. PMID 23893490
- [Background] Persson J, Hasselstrom J, Maurset A, Oye I, Svensson JO, Almqvist O, Scheinin H, Gustafsson LL, Almqvist O. Pharmacokinetics and non-analgesic effects of S- and R-ketamines in healthy volunteers with normal and reduced metabolic capacity. Eur J Clin Pharmacol. 2002 Feb;57(12):869-75. doi: 10.1007/s002280100353. PMID 11936706
- [Background] Sapkota A, Khurshid H, Qureshi IA, Jahan N, Went TR, Sultan W, Alfonso M. Efficacy and Safety of Intranasal Esketamine in Treatment-Resistant Depression in Adults: A Systematic Review. Cureus. 2021 Aug 21;13(8):e17352. doi: 10.7759/cureus.17352. eCollection 2021 Aug. PMID 34447651
- [Background] Bornemann-Cimenti H, Wejbora M, Michaeli K, Edler A, Sandner-Kiesling A. The effects of minimal-dose versus low-dose S-ketamine on opioid consumption, hyperalgesia, and postoperative delirium: a triple-blinded, randomized, active- and placebo-controlled clinical trial. Minerva Anestesiol. 2016 Oct;82(10):1069-1076. Epub 2016 Jun 21. PMID 27327855
- [Background] Hu ZC, Xu G, Zhang XW, Ma K, Jin JJ, Li PS. [Meta-analysis of the effects of dexmedetomidine combined with ketamine during dressing changes in burn patients]. Zhonghua Shao Shang Za Zhi. 2020 Jun 20;36(6):458-464. doi: 10.3760/cma.j.cn501120-20190327-00145. Chinese. PMID 32594705
- [Background] Lee KH, Lee SJ, Park JH, Kim SH, Lee H, Oh DS, Kim YH, Park YH, Kim H, Lee SE. Analgesia for spinal anesthesia positioning in elderly patients with proximal femoral fractures: Dexmedetomidine-ketamine versus dexmedetomidine-fentanyl. Medicine (Baltimore). 2020 May;99(20):e20001. doi: 10.1097/MD.0000000000020001. PMID 32443302
- [Background] Huge V, Lauchart M, Magerl W, Schelling G, Beyer A, Thieme D, Azad SC. Effects of low-dose intranasal (S)-ketamine in patients with neuropathic pain. Eur J Pain. 2010 Apr;14(4):387-94. doi: 10.1016/j.ejpain.2009.08.002. Epub 2009 Sep 3. PMID 19733106
- [Background] Chen LX, Ji DH, Zhang F, Li JH, Cui L, Bai CJ, Liu H, Liang Y. Richards-Campbell sleep questionnaire: psychometric properties of Chinese critically ill patients. Nurs Crit Care. 2019 Nov;24(6):362-368. doi: 10.1111/nicc.12357. Epub 2018 Jul 30. PMID 30062842
- [Background] Schug SA, Lavand'homme P, Barke A, Korwisi B, Rief W, Treede RD; IASP Taskforce for the Classification of Chronic Pain. The IASP classification of chronic pain for ICD-11: chronic postsurgical or posttraumatic pain. Pain. 2019 Jan;160(1):45-52. doi: 10.1097/j.pain.0000000000001413. PMID 30586070
- [Background] Werner MU, Kongsgaard UE. I. Defining persistent post-surgical pain: is an update required? Br J Anaesth. 2014 Jul;113(1):1-4. doi: 10.1093/bja/aeu012. Epub 2014 Feb 18. No abstract available. PMID 24554546